CLINICAL TRIAL: NCT05065112
Title: Individualised MApping-Guided Ablation to Improve Outcomes in pErsistent Atrial Fibrillation
Brief Title: Individualised Mapping in Persistent AF Ablation
Acronym: IMAGE AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 297733
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; catheter ablation; individualized mapping; focal activity; rotational activity
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI only (Active Comparator): Patients in this arm will undergo only standard pulmonary veins isolation with radiofrequency (RF) energy to treat their AF.
  Interventions: Procedure: Pulmonary veins isolation
- PVI + IM (Experimental): Patients in this arm will undergo standard wide area circumferential pulmonary veins isolation along with radiofrequency energy and additional RF ablation guided by individualised mapping with Cartofinder to treat their AF.
  Interventions: Procedure: Pulmonary veins isolation + Cartofinder-guided ablation

INTERVENTIONS:
Procedure: Pulmonary veins isolation + Cartofinder-guided ablation — The individualised mapping with Cartofinder intends to identify areas with the repetitive atrial activation patterns which are targeted with focal or linear ablation anchored on at least one end in an anatomical or electrical barrier.
  Arms: PVI + IM
Procedure: Pulmonary veins isolation — Wide area circumferential pulmonary veins isolation
  Arms: PVI only

SUMMARY:
A clinical randomised trial to compare strategies for ablation in persistent and long-standing persistent atrial fibrillation comprising of two arms: pulmonary veins isolation (PVI) only and PVI + individualised mapping-guided ablation (Cartofinder, Biosense Webster Inc.)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Signed informed consent.
3. Scheduled to undergo a clinically indicated, first-time catheter ablation procedure for the treatment of persistent atrial fibrillation.
4. In atrial fibrillation at the time of the index procedure.

Exclusion Criteria:

1. Paroxysmal atrial fibrillation.
2. Previous ablation procedure for atrial fibrillation.
3. Left ventricular ejection fraction < 45%
4. Obesity with BMI > 35 kg/m2
5. Congenital heart disease.
6. Previous cardiac surgery with atriotomy.
7. Previous left atrial appendage closure/ligation.
8. Contraindications to systemic anticoagulation, catheter ablation, and/or general anaesthesia.
9. Pregnancy
10. Current enrolment in a study evaluating another device or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia | 12 monts
  Freedom from any atrial arrhythmia without the use of antiarrhythmic drugs

SECONDARY OUTCOMES:
Freedom from atrial fibrillation | 12 months
  Freedom from atrial fibrillation without the use of antiarrhythmic drugs
Atrial fibrillation burden reduction | 12 months
  Reduction of the atrial fibrillation burden by 75% compared to baseline
Absolute atrial fibrillation burden | 12 months
  Absolute atrial fibrillation burden after a single, first-time ablative procedure guided by individualised mapping vs. standard approach.

CONTACTS AND LOCATIONS:
Overall Officials: Vias Markides, MD, FESC, Study Director — Royal Brompton Hospital, London, UK

IPD SHARING:
Plan to Share IPD: No